CLINICAL TRIAL: NCT05732077
Title: Fractional Flow Reserve to Determine the ApproprIateness of Percutaneous Renal Artery Intervention in Atherosclerosis Renovascular Hypertension Patients: a Pilot Randomized Trial
Brief Title: Fractional Flow Reserve to Determine Atherosclerosis Renovascular Hypertension Stenting
Acronym: FAIR-Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jianping LI, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022CR77
Record Dates: First submitted 2023-01-27; First posted 2023-02-16 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Renal Artery Stenosis Atherosclerotic; Secondary Hypertension Renal Arterial
MeSH Terms: interventions — Dopamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Not stenting (Other): Hyperemic FFR induced by 50μg/kg of dopamine via renal artery will be measured. If FFR is ≥0.80, randomization will be applied, and no stenting will be implanted. If FFR is <0.80, randomization will be ignored, and stenting will be performed.
  Interventions: Drug: Dopamine; Diagnostic Test: Fractional Flow Reserve, Renal; Device: Renal artery stenting
- Stenting (Other): Hyperemic FFR induced by 50μg/kg of dopamine via renal artery will be measured. No matter FFR is, stenting will be performed as planned.
  Interventions: Drug: Dopamine; Diagnostic Test: Fractional Flow Reserve, Renal; Device: Renal artery stenting

INTERVENTIONS:
Drug: Dopamine — A bolus dose of 50μg/kg dopamine via renal artery to induce hyperemic status
Diagnostic Test: Fractional Flow Reserve, Renal — Renal FFR will be measured based on SOP
Device: Renal artery stenting — Renal artery stenting will be implanted based on the protocol

SUMMARY:
Although randomized trials have demonstrated there is no benefit of renal-artery stenting in addition to medical therapy for patients with atherosclerosis renal artery stenosis, many patients indeed gained benefit in daily practices after stenting, such as reduction in blood pressure and recovery in renal functions. One important gap is that there is no universal standard to determine whether to stent in these patients. Fraction Flow Reserve (FFR) has been studied for many year in chronic coronary heart disease and FFR-guided revascularization strategy is known to be better than both angiography-guided revascularization and medication alone. The goal of this clinical trial is to learn whether Fraction Flow Reserve (FFR) is appropriate to determine stenting in hypertension patients with atherosclerosis renal artery stenosis. The main questions it aims to answer are:

* Is it appropriate to use FFR to determine whether or not stenting for hypertension patients with atherosclerosis renal artery stenosis?
* To provide detailed data supporting design of further trial, such as sample size calculating, cut-off value for FFR in renal artery stenosis, etc.

Participants met the inclusive/exclusive criteria will be randomized to stenting or not in the renal artery, then hyperemic FFR induced by dopamine will be measured in all participants. If FFR is ≥0.80, randomization will be applied. If FFR is <0.80, randomization will be ignored, and stenting will be performed as planned. The blood pressure and anti-hypertensive medications will be compared before and 3 months after the procedure based on ambulatory blood pressure monitoring, all participants will be followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* With recorded hypertension, AND the blood pressure is not controlled (SBP ≥140mmHg and/or DBP ≥90mmHg) on 2 or more classes of anti-hypertensive drugs;
* Evidence of renal artery stenosis and undergoing renal artery angiography;
* Able to follow the study protocol and provide informed consent;
* Renal artery angiography shows at least 1 main artery with stenosis of 50%-90%, AND the diameter is ≥ 4.0mm.

Exclusion Criteria:

* SBP ≥200mmHg and/or DBP ≥120mmHg at the day or randomization;
* Fibromuscular dysplasia or other non-atherosclerotic renal artery stenosis;
* Pregnancy or unknow pregnancy status in female of childbearing potential;
* Participation in any drug or device trial during the study period;
* Any stroke/TIA, OR with ≥70% stenosis of carotid artery;
* Any major surgery, myocardial infarction or interventional therapy 30 days prior to study entry;
* LVEF <30%;
* Comorbid condition causing life expectancy ≤1 year;
* Allergy to contrast or any of the following: aspirin, clopidogrel;
* Previous kidney transplant;
* Previous renal artery bypass surgery or stent intervention;
* Kidney size less than 8 cm measured by ultrasound;
* Local lab serum Cr >3.0 mg/dl (265.2μmol/l) on the day of randomization;
* Reference vessel size <4 mm or >8 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in daytime mean systolic blood pressure as measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM) | From baseline to 3 months post-procedure
Change in the composite index of antihypertensive drugs | From baseline to 3 months post-procedure
  Change in the composite index of antihypertensive drugs. Drug Composite Index = Weight (number of classes of antihypertensive drugs) × (sum of doses)

SECONDARY OUTCOMES:
Change in systolic blood pressure as measured by 24-hour ABPM | From baseline to 3 months post-procedure
Change in diastolic blood pressure as measured by 24-hour ABPM | From baseline to 3 months post-procedure
Change in home blood pressure | From baseline to 3 months post-procedure
Change in office blood pressure | From baseline to 3 months post-procedure
Change in the composite index of antihypertensive drugs to reach target blood pressure | From baseline to 1 year post-procedure
  Change in the composite index of antihypertensive drugs to reach target blood pressure. Drug Composite Index = Weight (number of classes of antihypertensive drugs) × (sum of doses)
Change in ABPM | From baseline to 6 months, 1 year post-procedure
All-cause death | From baseline to 1 year post-procedure
Cardiac death | From baseline to 1 year post-procedure
Acute myocardial infarction incidence | From baseline to 1 year post-procedure
  Based on universal definition of acute myocardial infarction
Non-fatal stroke incidence | From baseline to 1 year post-procedure
  Based on medical records under outcome committee's judge
Rehospitalization due to heart failure incidence | From baseline to 1 year post-procedure
  Based on medical records under outcome committee's judge
Increase in serum creatinine or dialysis | From baseline to 1 year post-procedure

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Chao-yang hospital, capital medical university, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qinghai province cardiovascular and cerebrovascular disease specialist hospital, Xining, Qinghai
  - Zibo Central Hospital, Zibo, Shandong
  - Peking University First Hospital Taiyuan Hospital, Taiyuan, Shanxi
  - Tianjin Beichen Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Li Y, Zheng J, Lu C, Fan F, Liu Z, Liu S, Yi T, Zhang L, Weng H, Wang B, Liu X, Zhou H, Ma D, Jia Z, Xiang L, Yang R, Shi D, Chen H, Xu L, Liu C, Kario K, Zhang Y, Li J. Fractional flow reserve-guided renal artery stenting in atherosclerotic renovascular hypertension: the FAIR randomized trial. Eur Heart J. 2025 Oct 7:ehaf746. doi: 10.1093/eurheartj/ehaf746. Online ahead of print. PMID 41056188